CLINICAL TRIAL: NCT04104022
Title: Treating Posttraumatic Stress Disorder in Patients With Opioid Use Disorder
Brief Title: Prolonged Exposure Therapy for PTSD and Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Kelly Peck, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRBSS #STUDY00000318; P20GM103644 (NIH)
Record Dates: First submitted 2019-09-17; First posted 2019-09-26 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Post Traumatic Stress Disorder; Opioid-use Disorder
Keywords: Post Traumatic Stress Disorder; Opioid-use Disorder; Prolonged Exposure Therapy; Opioid Agonist Therapy; Financial Incentives; Substance Use
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The present study is a three condition, parallel group, randomized trial to investigate the contribution of prolonged exposure therapy (PET) above and beyond opioid agonist treatment (OAT) alone for reducing PTSD symptoms among adults with concurrent PTSD and opioid use disorder. Participants will be randomized to one of three conditions: (a) OAT as usual, (b) OAT+PET, or (c) OAT+Enhanced PET (OAT+PET+). Those randomized to OAT as usual will continue to receive standard buprenorphine or methadone treatment from their current treatment provider and complete assessments of PTSD symptom severity, psychosocial functioning and drug use at intake and Study Weeks 4, 8, and 12. In addition to receiving OAT and completing monthly assessments, OAT+PET participants will receive 12 weekly PET sessions with a trained therapist. Finally, OAT+PET+ participants will receive the procedures for the OAT+PET group plus monetary incentives contingent upon completion of PET sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OAT as usual (No Intervention): Those randomized to OAT as usual will continue to receive standard buprenorphine or methadone treatment and complete assessments of PTSD symptom severity, psychosocial functioning and drug use at intake and Study Weeks 4, 8, and 12.
- OAT+PET (Active Comparator): In addition to receiving OAT and completing monthly assessments, OAT+PET participants will receive 12 weekly PET sessions with a trained therapist.
  Interventions: Behavioral: Prolonged Exposure Therapy
- OAT+PET+ (Experimental): OAT+PET+ participants will receive the procedures for the OAT+PET group plus monetary incentives contingent upon completion of PET sessions
  Interventions: Behavioral: Prolonged Exposure Therapy; Behavioral: Attendance-based monetary incentives

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — Within the general population, prolonged exposure therapy (PET) is a widely-used, empirically-supported and manualized therapy that is regarded as a first-line cognitive-behavioral treatment for posttraumatic stress disorder (PTSD). PET is designed to disrupt the cycle of anxiety and avoidance that characterizes PTSD via sustained imaginal and in-vivo exposure exercises that deliberately and systematically expose patients to painful memories and current, real-life trauma reminders that were previously avoided, yet not inherently harmful. Overall, PET has well-documented efficacy for reducing PTSD symptom severity in both civilian and veteran populations. PET is effective for reducing PTSD symptoms regardless of whether it is delivered remotely or face-to-face. Recent data also suggest that PET can improve PTSD symptoms without exacerbating substance use or craving among patients with substance use disorders when PET and substance use disorder treatment are delivered concurrently.
  Arms: OAT+PET; OAT+PET+
Behavioral: Attendance-based monetary incentives — Participants will earn vouchers that have monetary value for attending scheduled PET appointments. Each consecutive attended session will increase the voucher amount so that each consecutively attended appointment is worth an incrementally higher dollar amount. To support completion of the full 12-week PET protocol, we will also incorporate additional strategically-placed bonuses into the reinforcement schedule with the goal of maximizing the percentage of subjects who complete the full 12-session protocol. First, to support consistent (vs. sporadic) attendance, participants will receive a bonus for every two consecutive sessions attended. Second, to support completion of the full PET protocol, participants will receive an additional bonus upon completion of Session 12.
  Other Names: Contingency management
  Arms: OAT+PET+

SUMMARY:
Among patients with opioid use disorder (OUD), 90% report lifetime trauma exposure and 33% meet criteria for posttraumatic stress disorder (PTSD). The co-occurrence of OUD and PTSD is associated with worse mental health and opioid agonist treatment (OAT) outcomes relative to either diagnosis alone. Prolonged exposure therapy (PET) is an efficacious cognitive-behavioral treatment for reducing PTSD severity. Although preliminary findings indicate that PET may reduce PTSD symptom severity among patients receiving treatment for concomitant OUD, it is unclear to what extent improvements were a function of PET versus the effects of OAT itself. Therefore, the question of whether OAT alone may attenuate PTSD symptoms in the absence of intensive cognitive-behavioral therapy remains unanswered.

In this 12-week trial, we aim to investigate the contribution of PET above and beyond OAT alone for reducing PTSD symptoms among adults with concurrent PTSD and OUD. Participants will be randomized to one of three conditions: (a) OAT as usual, (b) OAT + PET, or (c) OAT + Enhanced PET (OAT+PET+). Those randomized to OAT as usual will continue to receive standard buprenorphine or methadone treatment from their current treatment provider and complete assessments of PTSD symptom severity, psychosocial functioning and drug use at intake and Study Weeks 4, 8, and 12. In addition to receiving OAT and completing monthly assessments, OAT+PET participants will receive PET consisting of 12 weekly, individual sessions with a trained therapist. Finally, OAT+PET+ participants will receive the procedures noted above for the OAT+PET group plus monetary incentives delivered contingent upon completion of PET sessions. Given the poor PET adherence rates reported among patients with substance use disorders, the use of incentives will ensure that we evaluate PET effects among patients who receive a sufficient dose of therapy. The proposed study design will permit us to disentangle the effects of PET from the effects of OAT alone while also including experimental conditions that reflect real-world practice. Taken together, this project will produce important new scientific and clinically-relevant information related to the mechanisms through which OAT and PET promote reductions in PTSD symptomatology in a highly vulnerable clinical population.

DETAILED DESCRIPTION:
Among patients with opioid use disorder (OUD), 90% report lifetime trauma exposure and 33% meet criteria for posttraumatic stress disorder (PTSD). The co-occurrence of OUD and PTSD is associated with more severe mental health symptoms and worse opioid agonist treatment (OAT) outcomes relative to either diagnosis alone. Prolonged exposure therapy (PET) is an efficacious manualized cognitive-behavioral treatment for reducing PTSD severity. Although preliminary findings indicate that PET may reduce PTSD symptom severity among patients receiving treatment for concomitant OUD, it is unclear to what extent observed improvements were a function of PET versus the psychopharmacological effects of OAT itself. Therefore, the question of whether OAT alone may attenuate PTSD symptomatology in the absence of intensive cognitive-behavioral therapy remains unanswered and is important given the prevalence and deleterious effects of PTSD among OAT patients, as well as the ever-present constraints on mental health resources in substance use treatment settings.

The present study will investigate the contribution of PET above and beyond OAT alone for reducing PTSD symptomatology among adults with concurrent PTSD and OUD. Eligible participants who complete the informed consent process will be randomized to one of three conditions: (a) OAT as usual, (b) OAT + PET, or (c) OAT + Enhanced PET (OAT+PET+). Those randomized to OAT as usual will continue to receive standard buprenorphine or methadone treatment from their current treatment provider and complete assessments of PTSD symptom severity, psychosocial functioning and drug use at intake and Study Weeks 4, 8, and 12. Follow-up assessment visits will be conducted in-person at our clinic following all relevant COVID-19-related CDC guidelines and university safety protocols. However, study measures may also be administered remotely via phone or telemedicine to reduce the risk of COVID-19 transmission. In addition to receiving OAT and completing monthly assessments, OAT+PET participants will receive PET consisting of 12 weekly, individual sessions with a trained therapist. Therapy sessions will be conducted at our research clinic or remotely via telemedicine to reduce the risk of COVID-19 transmission. Finally, OAT+PET+ participants will receive the procedures noted above for the OAT+PET group plus monetary incentives delivered contingent upon completion of PET sessions. Given the poor PET adherence rates reported among patients with substance use disorder (SUDs), the use of incentives will ensure that we evaluate PET effects among patients who receive a sufficient dose of therapy.

For inclusion in the study, participants must meet the following criteria: (a) > 18 years of age, (b) currently maintained on a stable methadone or buprenorphine dose for the treatment of OUD for >1 month prior to the study, (c) endorse >1 lifetime traumatic event, and (c) meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) PTSD diagnostic criteria (American Psychiatric Association, 2013). Exclusion criteria include: (a) the presence of an acute psychotic disorder, bipolar disorder with an active manic episode (but not simply the presence of bipolar disorder), (b) imminent risk for suicide, (c) a medical condition that may interfere with consent or participation (e.g., organic brain syndrome, dementia, head injury, neuropathy, etc.), and (d) illiteracy in English.

Participants randomized to OAT as usual will continue to receive standard buprenorphine or methadone maintenance from their current treatment provider and complete assessments of PTSD symptom severity, psychosocial functioning and drug use at Study Weeks 4, 8, and 12. Follow-up assessment visits will be conducted in-person at our clinic following all relevant COVID-19-related CDC guidelines and university safety protocols. However, study measures may also be administered remotely via phone or telemedicine to reduce the risk of COVID-19 transmission. In addition to receiving standard buprenorphine- or methadone-maintenance treatment as described above and completing monthly assessments, OAT+PET participants will also receive 12 individual sessions of PET. Therapy sessions will be conducted at our research clinic or remotely via telemedicine to reduce the risk of COVID-19 transmission. Beginning in Study Week 1, OAT+PET participants will complete weekly 60-minute PET sessions provided by a therapist trained in PET. Participants randomized to the OAT+PET+ condition will receive the procedures noted above for the OAT+PET group plus monetary incentives delivered contingent upon completion of PET sessions. Each consecutive attended session will increase the voucher amount so that each consecutively attended appointment is worth an incrementally higher dollar amount. To support completion of the full 12-week PET protocol, we will also incorporate additional strategically-placed bonuses into the reinforcement schedule with the goal of maximizing the percentage of subjects who complete the full 12-session protocol. First, to support consistent (vs. sporadic) attendance, participants will receive a bonus for every two consecutive sessions attended. Second, to support completion of the full PET protocol, participants will receive an additional bonus upon completion of Session 12.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* currently maintained on a stable methadone or buprenorphine dose for >1 month prior to the study
* endorse >1 lifetime traumatic event
* meet current DSM-V posttraumatic stress disorder criteria

Exclusion Criteria:

* Presence of an acute psychotic disorder, bipolar disorder with an active manic episode
* imminent risk for suicide
* a medical condition that may interfere with consent or participation
* illiteracy in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Peck, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vemont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peck KR, Giannini J, Badger GJ, Cole R, Sigmon SC. A novel prolonged exposure therapy protocol for improving therapy session attendance and PTSD symptoms among adults receiving buprenorphine or methadone treatment. Drug Alcohol Depend. 2025 Jan 1;266:112507. doi: 10.1016/j.drugalcdep.2024.112507. Epub 2024 Nov 27. PMID 39642783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Started | 17 | 17 | 18
Completed | 17 | 12 | 18
Not Completed | 0 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+ | Total
Number analyzed (Participants) | 17 | 17 | 18 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (10.8) | 39.9 (10.2) | 37.2 (10.8) | 39.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 13 | 36
  Male | 5 | 6 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 15 | 15 | 17 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 15 | 15 | 17 | 47
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 18 | 52
Medication Use to Treat Opioid Use Disorder [Count of Participants; unit: Participants]
  Buprenorphine | 12 | 12 | 11 | 35
  Methadone | 5 | 5 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Posttraumatic Stress Disorder (PTSD) Symptom Severity
Description: Change in PTSD symptom severity will be measured by the total symptom severity score of the Clinician Administered PTSD Scale for DSM-V (CAPS-5). The CAPS-5 is a clinician-administered clinical interview that produces a total symptom severity score that is obtained by summing the scores for each of the 20 items. Scores range from 0-80 with lower scores indicating less severe symptoms of PTSD. A negative sign in front of a number represents a decrease in score and less severe PTSD symptoms at 12 weeks compared to baseline. A greater decrease in score represents greater reduction in symptoms (more positive outcomes).
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 17 | 17 | 18
Score on a scale | -11.4 (2.7) | -12.8 (3.1) | -18.3 (2.6)

2. Secondary Outcome: Posttraumatic Stress Disorder (PTSD) Symptom Severity
Description: Mean PTSD symptom severity will be measured by the PTSD Checklist for DSM-V (PCL-5) total score. The PCL-5 is a self-report measure that produces a total score that is obtained by summing the scores for each of the the 20 items. Scores range from 0-80 with higher scores indicating more severe symptoms of PTSD.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 17 | 17 | 18
Score on a scale | 31.8 (3.7) | 28.9 (4.4) | 21.7 (3.5)

3. Secondary Outcome: Anxiety Symptom Severity
Description: Mean anxiety symptom severity will be measured by the Beck Anxiety Inventory (BAI) total score. The BAI is a self-report measure that produces a total score that is obtained by summing the scores for each of the 21 items. Scores range from 0-63 with higher scores indicating more severe symptoms of anxiety.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 17 | 17 | 18
Score on a scale | 18.1 (2.6) | 15.2 (3.0) | 13.9 (2.5)

4. Secondary Outcome: Depression Symptom Severity
Description: Mean depression symptom severity will be measured by the Beck Depression Inventory (BDI-II) total score. The BDI-II is a self-report measure that produces a total score that is obtained by summing the scores for each of the 21 items. Scores range from 0-63 with higher scores indicating more severe symptoms of depression.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 17 | 17 | 18
Score on a scale | 22.4 (3.0) | 23.1 (3.3) | 18.6 (2.8)

5. Secondary Outcome: Number of Participants Achieving Illicit Opioid Abstinence
Description: Illicit opioid abstinence will be measured by the overall percentage of urinalyses biochemically verified to be abstinent for illicit opioids at the end of the intervention period.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 15 | 10 | 15
Participants | 13 | 8 | 14

6. Secondary Outcome: Psychiatric Problems Related to Substance Use
Description: Psychiatric problems related to substance use will be measured by the Addiction Severity Index (ASI) Psychiatric subscale score. The ASI is a clinician-administered structured interview. Scores for this subscale range from 0-1 with higher scores indicating more severe psychiatric consequences of substance use.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 17 | 17 | 18
Score on a scale | 0.39 (0.04) | 0.37 (0.05) | 0.33 (0.04)

7. Secondary Outcome: Number of Participants Who Report Abstinence From Illicit Non-opioid Substance Use
Description: Abstinence from illicit non-opioid substance use will be measured by the Timeline Follow-back (TLFB). The TLFB will be administered by an interviewer and involves participants retrospectively estimating their illicit non-opioid substance use (e.g., amphetamines, benzodiazepines, cocaine) during the 30 days prior to the interview date. Abstinence from illicit non-opioid substance use will be measured by the overall number of participants reporting abstinence from illicit non-opioid substances .
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 15 | 10 | 13
Participants | 11 | 8 | 13

8. Secondary Outcome: Pain Intensity and Interference
Description: For participants who endorsed the presence of pain during the past month, pain intensity and interference will be measured by Brief Pain Inventory -Short Form (BPI-SF). The BPI-SF is a self-report measure of pain intensity and interference in function during the past week. The pain intensity section of the BPI includes a rating of average pain intensity; whereas, the functional interference section consists of a rating of pain interference on general activity. Items assessing pain intensity and functional interference are scored from 0-10 with higher scores indicating greater pain severity and functional interference, respectively.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 9 | 3 | 6
Score on a scale
  Pain intensity | 4.9 (2.6) | 5.0 (2.0) | 4.0 (2.4)
  Pain interference | 6.0 (3.6) | 5.0 (4.4) | 5.8 (2.2)

9. Secondary Outcome: Delay Discounting
Description: Rates of delay discounting will be measured by the Monetary Choice Questionnaire (MCQ). The MCQ is a 27-item self-report measure consisting of items that presents a choice between smaller, immediate and larger, delayed monetary rewards. Immediate reward values ranged from $11 to $80, delayed rewards ranged from $25 to $85 and the length of the delay ranged from 7 days to 186 days. "Discounting rates," or k-values, are calculated from individuals' choices across items and represent rates at which the individual devalues rewards overall. The estimate of participant's discounting "k" was estimated with the following formula: V = A/(1+kD) where V is the present discounted value of the reinforcer, A is the objective value of the reinforcer, D is the delay until the receipt of the reinforcer, and k is the derived parameter that corresponds to the rate of discounting. In this equation, larger k values correspond to greater discounting of delayed rewards, or preference for small
Time Frame: 12 weeks
Measure: Geometric Mean (Standard Error); unit: K-Value
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 16 | 17 | 17
K-Value | 0.05 (0.02) | 0.02 (0.01) | 0.03 (0.01)

10. Secondary Outcome: Insomnia Severity
Description: Insomnia severity will be measured by the Insomnia Severity Index (ISI). The ISI is a self-report measure that consists of 7 items that are scored from 0-4. The ISI produces a total score that is obtained by summing the scores for each of the the 7 items. Scores range from 0-28 with higher scores indicating more severe symptoms of insomnia.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
Number analyzed (Participants) | 17 | 17 | 18
Score on a scale | 15.0 (1.6) | 14.7 (1.9) | 13.0 (1.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | OAT as Usual | OAT+PET | OAT+PET+
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 4/17 | 2/17 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OAT as Usual (N=17) | OAT+PET (N=17) | OAT+PET+ (N=18)
Adverse events not categorized by organ system (General disorders) | 4 (5) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT04104022/Prot_SAP_000.pdf